CLINICAL TRIAL: NCT05304988
Title: Development and Validation of the Exercise Fit Test (EFT) for Adolescents With Cancer
Brief Title: Development and Validation of the EFT for Adolescents With Cancer
Status: Recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Katherine Lam, Assistant Professor, The Hong Kong Polytechnic University
Other Study IDs: EFT_Adolescents
Record Dates: First submitted 2021-05-18; First posted 2022-03-31 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: Adolescents; Physical Activity; Tool
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Developing and testing of EFT: It aims to develop a patient-based assessment tool by our research members for adolescents with cancer in Hong Kong.
  Interventions: Other: Testing of the EFT

INTERVENTIONS:
Other: Testing of the EFT — Our team will develop specific questions in EFT. Then, subject will be invited to fill in a set of questionnaires covering demographic characteristics, EFT items and a numerical rating scale for pain scores. The physiotherapists will rate the subject with the most appropriate level of physical activity.

SUMMARY:
There is increasing evidence of interventions shown to be effective to promote physical activity in adolescents with cancer. Nevertheless, adolescents with cancer become physically inactive after the end of the interventions. These interventions emphasized heavily on interventionists' role to assess adolescents' physical fitness and prescribe exercises. After the intervention, the adolescents were unable to follow the previous exercise prescriptions due to their changing medical conditions. To promote physical activity sustainably, it is vital to develop a patient-based assessment tool to allow adolescents with cancer to self-assess their own appropriate levels of physical activity that they could perform. However, a review of literature indicates a lack of such a tool.

DETAILED DESCRIPTION:
A cross-sectional study design will be used. A convenience sample of 400 adolescents who (1) are aged 13-18; (2) are diagnosed with cancer; (3) can communicate in Cantonese and read Chinese will be recruited in Hong Kong Children's Hospital. The outcome measures will include demographic characteristics, pain scores, cardiopulmonary function measurements, EFT scores and ratings of the physiotherapists for the fitness of subjects for physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13-18
* are diagnosed with cancer
* are able to communicate in Cantonese and read Chinese

Exclusion Criteria:

Those with physical or cognitive impairments and learning problems, as identified from the medical records, were excluded. Also, those with medical advice that physical activity was not recommended or with detailed exercise prescriptions from physicians or physiotherapists during recruitment were excluded.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A convenience sample of 400 adolescents who meet the eligibility criteria will be invited to participate. Subjects will be recruited in non-governmental organizations and Hong Kong Children's Hospital which is the largest hospital in Hong Kong for admitting adolescents with cancer for hospitalization and follow-ups.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The EFT scores | Just before their scheduled physiotherapists interview
  Subjects will be asked to mark their responses for the EFT items in the second draft just before their scheduled oncologist routine visit. The scale ranges from 1 to 5. Higher scores indicate that the subjects are fit for a higher level of physical activity.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) for pain | Just before their scheduled oncologist routine visit
  Subjects will be asked to mark their pain level on the NRS according to their experience just before their scheduled oncologist routine visit. The scale ranges from 0 to 10. Higher scores represent a higher level of pain.
The physiotherapists' rating for physical activity | Just before their scheduled physiotherapist interview
  The physiotherapists will rate the subject with the most appropriate intensity level of physical activity on a 5-point scale. The scale ranges from 1 to 5. Higher scores indicate that the subjects are fit for a higher level of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Lam, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Katherine Lam, Hong Kong, Hong Kong,China, Hong Kong

IPD SHARING:
Plan to Share IPD: No